CLINICAL TRIAL: NCT06971575
Title: Cervical Radiculopathy Imaging Using MR Neurography With Electrodiagnostic Correlation
Brief Title: Cervical Radiculopathy Imaging Using MRN With Electrodiagnostic Correlation
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1447
Record Dates: First submitted 2025-03-24; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cervical Radiculopathy Patients: Patients diagnosed with unilateral cervical radiculopathy and signs of clinical weakness.
  Interventions: Diagnostic Test: Magnetic resonance neurography

INTERVENTIONS:
Diagnostic Test: Magnetic resonance neurography — Patients will undergo a cervical MRI with specialized magnetic resonance neurography sequences to evaluate the extraforaminal cervical nerve roots.

SUMMARY:
This project will study patients with cervical radiculopathy. We will evaluate the combined diagnostic and prognostic value of magnetic resonance neurography (MRN), electrodiagnostic (EDX) studies, and historical and physical clinical elements. Specifically, this project will explore whether these data individually or in combination correlate with response to procedural and non-procedural treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with symptoms compatible with acute or subacute unilateral (one-sided) cervical radiculopathy and signs of clinical weakness
* 18-60 years old at the time of evaluation
* Symptom onset of 2 to 12 weeks leading up to baseline visit
* Diagnosis of unilateral cervical radiculopathy, with or without spinal cord compression, based on signs and symptoms, physical exam and supported by MRI findings of radiculopathy (as evidenced by foraminal stenosis/narrowing) based on standard-of-care cervical spine MRI
* Patients who have undergone or have planned electrodiagnostic testing at HSS prior to surgery

Exclusion Criteria:

* Prior cervical surgery or instrumentation
* Those who have had a prior episode of cervical radiculopathy
* History of peripheral neuropathy or another acute or chronic neurodegenerative condition
* History of stroke, cerebellar disease, or central nervous system disease
* Contraindications to undergoing a standard MRI examination (e.g., pregnancy)
* Patients presenting with bilateral cervical radiculopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with acute or subacute unilateral cervical radiculopathy and signs of clinical weakness
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Presence of abnormalities on nerve (MRN) imaging | Baseline
  Presence of abnormalities on cervical MRN imaging that correspond to clinical findings of cervical radiculopathy. This includes abnormalities in extraforaminal cervical nerve root intraneural T2 signal and DTI values.
Relationship between abnormalities on imaging and electrodiagnostic assessment | Baseline
  The relationship between any abnormalities identified on nerve imaging (cervical MRN) and electrodiagnostic findings will be assessed.

SECONDARY OUTCOMES:
Numeric rating scale (NRS) pain | Baseline, 3 months, 6 months, 12 months
  Current NRS pain will be assessed on 0-10 scales (10=worst pain).
Neck Disability Index (NDI) | Baseline, 3 months, 6 months, 12 months
  NDI is scored on a 0-100% scale, with 100% representing complete disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No